CLINICAL TRIAL: NCT07094035
Title: Efficacy Study of a Food Supplement Based on an Extract of Green Tea (Camellia Sinensis (L.) Kuntze - Folium) and a Pool of Probiotics (L. Plantarum, L. Rhamnosus and B. Animalis Subsp. Lactis) for the Management of Gastrointestinal Discomfort and for the Maintenance of the Balance of Intestinal Function in Subjects With Irritable Bowel Syndrome (Irritable Bowel Syndrome - IBS) With Predominance of Constipation (IBS-C): Single-center, Controlled, Randomized, Parallel-arm, Double-blind Clinical Trial.
Brief Title: The Beneficial Effects on the Intestinal Function of a Food Supplement Based on an Extract of Green Tea and a Pool of Probiotics in Subjects With Irritable Bowel Syndrome With Predominance of Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adamas Biotech S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IBS-THE-PROB25
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: IBS, Constipation Predominant
Keywords: IBS, constipation predominant; Food Supplement; Green tea extract; probiotics
MeSH Terms: conditions — Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1: active group who will take verum (Experimental): Subjects who will take the food supplement. The daily consumption of the food supplement provides: green tea extract (Camellia sinensis (L.) Kuntze - folium) 300 mg, as a green capsule, and a pool of probiotics (Lactobacillus rhamnosus LRH020 2x10^9 UFC, Bifidobacterium lactis BL050 2x10^9 UFC, Lactobacillus plantarum PBS067 2x10^9 UFC), as a white capsule.
  Interventions: Dietary Supplement: food supplement based on a mixture of green tea extract and a pool of probiotics.
- GROUP 2: subjects who will take PLACEBO (Placebo Comparator): Subjects who will take daily: 1 capsule/day of maltodextrin (500 mg) with a green shell, and 1 capsule/day of maltodextrin (500 mg) with a white shell for 56 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: food supplement based on a mixture of green tea extract and a pool of probiotics. — two capsules of food supplement (verum) or placebo, daily for 56 consecutive days. The daily consumption of the food supplement provides: green tea extract (Camellia sinensis (L.) Kuntze - folium) 300 mg, as a green capsule, and a pool of probiotics (Lactobacillus rhamnosus LRH020 2x10^9 UFC, Bifidobacterium lactis BL050 2x10^9 UFC, Lactobacillus plantarum PBS067 2x10^9 UFC), as a white capsule.
  Arms: GROUP 1: active group who will take verum
Dietary Supplement: Placebo — 1 capsule/day of maltodextrin (500 mg) with a green shell, and 1 capsule/day of maltodextrin (500 mg) with a white shell for 56 days. The two colours are applied to maintain the binding.
  Arms: GROUP 2: subjects who will take PLACEBO

SUMMARY:
The study will aim to evaluate the effectiveness of the use of a food supplement, based on a green tea extract (Camellia sinensis (L.) Kuntze - folium) and a pool of probiotics (L. plantarum, L. rhamnosus and B. animalis subsp. lactis), in the management of gastrointestinal distress in the general population and in subjects with IBS in the predominant form of IBS-C, with an impact on quality of life.

The primary outcome is the overall improvement of perceived gastrointestinal symptoms in subjects with IBS in the predominant form of IBS-C; than the secondary outcomes are the 1) assessment of the impact of constipation on perceived quality of life in the last 4 weeks, 2) effectiveness in improving stool consistency, 3) effectiveness of the frequency of bowel movements, 4) efficacy with respect to the frequency and intensity of the characteristic symptoms of IBS, 5) effectiveness of the decrease in frequency in the use of salvage treatments 6) efficacy against abdominal pain to be evaluated separately from intestinal discomfort 7) evaluation of the reduction of intestinal inflammatory status through the analysis of fecal inflammatory markers Calprotectin and Zonulin and 8) probiotic colonization rate, improving the quality of life of the subjects affected by IBS-C.

DETAILED DESCRIPTION:
The IBS-THE-PROB25 study aims to understand whether a food supplement based on green tea and a mix of probiotics can help people suffering from Irritable Bowel Syndrome with constipation (IBS-C). The main goal is to see if this supplement improves the overall symptoms perceived by people with IBS-C.

Study participants are between 18 and 70 years old and have symptoms of IBS-C for at least 3 months, with constipation problems such as going to the bathroom less than 3 times a week and often having hard stools. There are also criteria why some people will not be able to participate, such as those who have other intestinal diseases or take certain medications.

Participants will be randomly divided into two groups. One group will take the supplement with green tea and probiotics, the other group will take a placebo (an inactive substance that looks the same as the supplements). In particular, the study plans to recruit 64 subjects (32 subjects per group), who will be randomized into the following experimental groups:

GROUP 1 (32 subjects) subjects who will have to take the food supplement, an extract of green tea (Camellia sinensis (L.) Kuntze - folium) and a pool of probiotics (L. plantarum, L. rhamnosus and B. animalis subsp. lactis) GROUP 2 (32 subjects) subjects who will have to take placebo. Each subject of the two experimental groups before, during and after the administration of the dietary supplement or placebo, will undergo the evaluation of the primary and secondary outcomes. Neither participants nor doctors will know who is taking what (double-blind study). Clinicians will collect information about participants symptoms through questionnaires.

Specifically, a questionnaire called IBS-SSS will be used to assess the overall severity of symptoms. Quality of life, stool consistency (using the Bristol Scale), frequency of bowel movements, frequency and intensity of specific symptoms such as bloating and pain, use of "rescue" medications (such as laxatives) and abdominal pain will also be taken into account. A small group of participants will also need to provide stool samples to analyze substances that indicate inflammation and to see if probiotics "colonize" the gut.

The data collected will be analyzed with statistical methods to compare the two groups and see if there are significant differences in symptoms.

The trial will be conducted at a single center: COMEGEN Soc. Coop. Sociale, located in Viale Maria Bakunin, 41 (Parco S. Paolo), 80126- Naples. The Principal Investigator of the study is Dr. Matteo Laringe, also affiliated with COMEGEN Soc. Coop. Social. Subjects enrolled in the study will be followed at this location for the duration of their participation.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 70 years
* able to understand and sign informed consent
* HIV negative test
* negative pregnancy test
* With IBS symptoms for at least 3 months (with onset at least 6 months earlier)
* recurrent abdominal pain at least 1 day a week, associated with two or more of the following criteria: associated with the act of defecation, associated with a change in the frequency of bowel movements, associated with a change in the shape of the stool (Rome IV diagnostic criteria)
* who have less than three BM/wk and at least one of the following conditions:

  * in more than 25%* of defecatory acts
  * lumpy or hard stools (BSFS type 1 or 2) in more than 25% of bowel movements
  * feeling of incomplete evacuation in more than 25% of defecations
  * feeling of anorectal obstruction/blockage in more than 25% of defecations
  * carry out manual manoeuvres to facilitate evacuation in more than 25% of defecations
* Able to understand and comply with the requirements of the protocol.

Exclusion Criteria:

* pregnancy
* lactation
* HIV positive
* do not meet inclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the food supplement in the overall improvement of perceived gastrointestinal symptoms. | [Time frame: baseline (t0), day 28 (t28d), day 56 (t56d), day 84 (t84d)]
  Validated questionnaire for self-assessment of the severity of global gastrointestinal symptomatology characterizing IBS, IBS Severity Scoring System (IBS-SSS). The questionnaire consists of 5 items referring to: abdominal pain, bowel dysfunction and general well-being. It is commonly used as an outcome measure in clinical efficacy trials, due to its high sensitivity following treatment. The total score obtained allows to determine the severity of global gastrointestinal symptoms, whether IBS-related symptoms are mild, moderate or severe and whether, following treatment, there is an improvement in global symptoms in the treated group compared to the placebo group.

SECONDARY OUTCOMES:
Assessment of the impact of constipation on perceived quality of life in the last 4 weeks | [Time frame: baseline (t0), day 28 (t28d), day 56 (t56d), day 84 (t84d)]
  Quality of Life Questionnaire (Short Form Health Survey-12 -SF-12) was developed in a multiyear study of patients with chronic conditions. It is a validated questionnaire widely used in clinical practice for self-assessment of quality of life against a generic disorder. The SF-12 questionnaire allows you to describe the health of a subject through two synthetic indices calculated on 12 questions. The index called Physical Component Summary (PCS), concerns the physical state, while the Mental Component Summary (MCS) index measures the mental state.
The effectiveness in improving stool consistency. | [Time frame: baseline (t0), day 28 (t28d), day 56 (t56d), day 84 (t84d)]
  Bristol Stool Form Scale (BSFS), a validated instrument that assesses stool consistency on a spectrum of seven types. Type 1 and 2 stools denote hard or lumpy stools, while type 6 and 7 stools are indicative of loose or watery stools. The stools that characterize subjects with intestinal hyperactivity are type 5, 6, 7. Stool consistency will be reported by the subject at visits and reported, during the study period, on the Bowel Function Diary.
The effectiveness of the frequency of bowel movements. | [Time frame: baseline (t0), day 28 (t28d), day 56 (t56d), day 84 (t84d)]
  Number of bowel movements/week (BM/WK) will be reported by the subject at the visits (average BM/week over the previous 4 weeks) and reported, during the study period, on the bowel function diary.
The efficacy with respect to the frequency and intensity of the characteristic symptoms of IBS. | [Time frame: baseline (t0), day 28 (t28d), day 56 (t56d), day 84 (t84d)]
  The assessment of the frequency and intensity characteristics of the subject with constipated IBS form (feeling of bloating, abdominal distension, feeling of fullness, abdominal pain, flatulence) will be determined through the compilation of a 5-point Likert scale (0 no discomfort - 5 maximum discomfort), present within the bowel function diary. Daily registration is useful to avoid the "recall" bias that could occur when filling out questionnaires at pre-arranged visits.
The effectiveness of the decrease in frequency in the use of salvage treatments. | [Time frame: baseline (t0), day 28 (t28d), day 56 (t56d), day 84 (t84d)]
  The evaluation of the frequency of use of salvage treatments, such as drugs for bowel function, laxatives or antispasmodics, will be recorded through the compilation of the bowel function diary.
The efficacy against abdominal pain to be evaluated separately from intestinal discomfort. | [Time frame: baseline (t0), day 28 (t28d), day 56 (t56d), day 84 (t84d)]
  Visual Analogue Scale (VAS). It is a self-assessment tool for pain, used for several purposes and in the assessment of general pain in patients accessing the emergency room. It consists of a 10 cm strip of paper, which at both ends has the two endpoints "no pain" and "worst pain I can imagine", the patient must mark the level of perceived pain on the strip.
Evaluation of the reduction of intestinal inflammatory status through the analysis of fecal inflammatory markers Calprotectin and Zonulin | [Time frame: baseline (t0), day 56 (t56g), day 84 (t84g)]
  Investigation carried out on stool samples. This analysis will be carried out on a pool of 30 subjects, 15 from the treatment group and 15 from the placebo group.
Probiotic colonization rate. | [Time frame: baseline (t0), day 56 (t56g), day 84 (t84g)]
  Relative abundance of microbial species presents in the treatment (L. plantarum, L. rhamnosus, and B. animalis subsp. lactis) to assess the colonization ability of the study treatment. Investigation carried out on stool samples. This analysis will be carried out on a pool of 30 subjects, 15 from the treatment group and 15 from the placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- COMEGEN Soc. Coop. Sociale, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No